CLINICAL TRIAL: NCT02099526
Title: Needs of Older Caregivers of Adults With Cancer In the First 2 Weeks Following Hospital Discharge
Brief Title: Older Cancer Caregiver Needs Post Hospital Discharge
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: The Reed Foundation, Ruth Landes Memorial Research Fund (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00051203
Record Dates: First submitted 2014-03-26; First posted 2014-03-31 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-01

CONDITIONS: Cancer Caregivers of Older Adults
Keywords: cancer; caregiver; caregiving; care give; elderly; older adults; unmet needs; post-discharge; cancer symptoms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The goals of the study are to investigate the needs of older (age 60+) caregivers caring for adults with cancer at 1-week and 2 weeks following hospital discharge and to explore strategies that may assist caregivers in their home caregiving needs. This study will explore how these needs vary based on caregiver spirituality and relationship with the care recipient.

The study will enroll cancer patients and their caregivers admitted to 9100 and 9300, which are the hematological and non-hematological malignancy units at Duke University Medical Center (DUMC) respectively. Results of this study will lay the groundwork for creating tailored interventions for caregivers that are compatible to their preferences and more responsive to their needs.

DETAILED DESCRIPTION:
Baseline demographic data about the caregiver and patient will be collected at patient beside prior to hospital discharge. Qualitative interviews will be conducted with the cancer caregivers in their home at 1-week after their loved one was discharged from the hospital, and at 2-weeks after discharge from the hospital. This study utilizes a qualitative descriptive design.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver must speak English
* Caregiver must be at least 60 years of age
* Patients must be 18 years of age or older & speak English
* Patients must have been admitted to either the 9100 or 9300 oncology unit for treatment of cancer, or treatment-related/cancer-related complications
* Patients must be discharged home to participate in the study

Exclusion Criteria:

* Dyads who received hospice referral prior to the care recipient's discharge
* Patient must not have any diagnosis of dementia in their medical records, or any cognitive impairment as assessed by hospital providers (physicians and nurses)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects include 30 informal caregivers and cancer patients dyads. Patients have been admitted to either the hematological malignancy unit, or the non-hematological malignancy unit for treatment of cancer, or treatment-related/cancer-related complications.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Unmet cancer caregiver needs | 1 week after patient discharge from hospital
  Explore the needs (e.g., psychosocial) of older adults caring for a loved one with cancer at home during the first and second weeks after hospital discharge, and determine how these needs vary by spirituality and relationship to the care recipient.
Caregiver strategies assisting in caregiving role | 1 week after patient discharge from hospital
  Identify the strategies used by older caregivers during the first and second weeks after hospital discharge, and determine how these strategies vary by spirituality and relationship to the care recipient.
Caregiver decision making in seeking assistance for cancer patient | 1 week after patient discharge from hospital
  Describe the preferences of support and assistance (e.g., family/friends) of older caregivers in caring for a loved one with cancer at home during the first and second weeks after hospital discharge, and determine how these preferences vary by spirituality and relationship to the care recipient.

SECONDARY OUTCOMES:
Caregiver needs and preferences vary with time | 2 weeks after patient discharge from the hospital
  Explore whether caregiver needs and preferences vary with time (1 week versus 2 weeks post hospital discharge).

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Hendrix, DNS, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States